CLINICAL TRIAL: NCT01408771
Title: "Swallow my Urine Back" : Inhibition of Detrusor Overactivity by Swallowing Maneuver
Status: Completed | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Kobi Stav, Assaf-Harofeh Medical Center
Other Study IDs: 35/11
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-07

CONDITIONS: Overactive Detrusor
Keywords: Urodynamics; Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to find out whether swallowing has an effect on the degree of urinary urgency and on the amplitude of detrusor contraction during filling cystometry in patients with detrusor overactivity (DO).

DETAILED DESCRIPTION:
Consecutive patients with DO will be included in this study. During urodynamics, the amplitude of the waves of DO will be documented and compared. At the beginning of the 2nd wave, patients will be asked to perform 5 repetitive swallows. Following each wave, patients will be asked to grade the severity of the urgency by a visual analogue scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

patients with DO in filling cystometry

* antimuscarinic medications were requested to stop for 7 days before the cystometry

Exclusion Criteria: none

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are sedignated for urodynamic study with overactive bladder symptoms
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kobi Stav, MD, Principal Investigator — Assaf Harofeh Medical Center, Zeriffin, Israel